# Georgia State University Department of Health Promotion and Behavior School of Public Health Informed Consent

Title: Testing the efficacy of a web-based program for college women

Principal Investigator: Dr. Laura F. Salazar

Sponsor: National Institute of Alcohol Abuse and Alcoholism

### I. Purpose:

The purpose of this study is to examine the effectiveness of a 3-hour web-based program for incoming female freshmen. A total of 750 participants (250 from your university) will be invited to take part in this study. You are invited to take part in this research study because you are:

- female
- a freshman
- 18 to 20 years old
- a full-time student at Georgia State University, Emory University or University of Georgia

This research study is an NIH-funded clinical trial. All NIH funded studies that qualify as clinical trials must be registered at clinicaltrials.gov within 21 days of enrolling participants. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law.

□ "Please check this box if you have read this section on the purpose of the research study."

#### II. Procedures:

Version Date: July 31, 2018

If you decide to take part, you will take part in an online study. Participating in this study calls for about 5.5 hours of your time over the next six months. The study will involve:

- Completing a 45-minute online survey
- viewing a 4-part web-based program at your own pace (total time of program = 3 hours)
- Completing a 10-minute survey following each of the 4 parts
- Completing a second 45-minute online survey 6 months later
- The online survey will be on personal information (age, race, ethnicity, etc.), attitudes, health behaviors, dating behaviors, experiences of sexual violence, and perceptions of risk.
- The brief 10-minute surveys will ask your opinion on the program content.
- You will be randomized to view one of two different web-based programs. Each program covers topics related to female freshmen's mental and physical health and safety.



| | study." |
|---|---|
| | Future Research chers will take out information that may identify you and may use your data for future ch. If we do this, we will not ask for any additional consent for you. |
| | "Please check this box if you have read this section on the risks of the research study." |
| when a questic will be trained | is the possibility that taking part in this study may cause you to be nervous or stressed answering some of the questions or viewing the program; you do not have to answer any ons you do not want to answer in the survey. Also, if you feel too anxious or stressed, you a provided with the Principal Investigator's phone number. If you need or want to talk to a therapist, you will be provided a toll-free 800-hotline number for you to call. You will be given local university resources for you to contact. |
| | "Please check this box if you have read this section on the risks of the research study." |
| issues how th | Benefits: udy is designed to benefit you directly by increasing your understanding of health-related and how to decrease your risk of negative experiences. Overall, we hope to learn about its web-based program can help others like you to have healthier lives and a positive experience. |
| | "Please check this box if you have read this section on the benefits of the research study." |
| | ternatives: ternative to taking part in this study is to not take part in the study. |
| | "Please check this box if you have read this section on the compensation of the research study." |
| giftcare<br>the 6-n | Compensation: ill receive a \$25 Amazon e-giftcard for completing the baseline survey, a \$40 Amazon e-d for completing all four 10-minute surveys, and a \$40 Amazon e-giftcard for completing nonth follow-up survey. Overall, participants can earn up to \$105 in Amazon giftcards for part in this study. |

Version Date: July 31, 2018

| | "Please check this box if you have read this section on the compensation of the research study." |
|---|---|
| You do | Voluntary Participation and Withdrawal: o not have to be in this study. If you decide to be in the study and change your mind, you ne right to drop out at any time. You may skip questions or stop participating at any time. ver you decide, you will not lose any benefits to which you are otherwise entitled. |
| | "Please check this box if you have read this section on voluntary participation and withdrawal of the research study." |
| X. | Confidentiality: |
| We wi | ll keep your records private to the extent allowed by law. The following people and |
| entities | s will have access to the information you provide: |
| | Dr. Laura Salazar and other members of the research team |
| | GSU Institutional Review Board |
| | Office for Human Research Protection (OHRP) |
| | National Institutes of Health |

We will use only a unique study I.D. number rather than your name or email address on all study records where we can. Your name and other facts that might point to you will not appear when we present this study or publish its results. In addition, we will make sure your information is kept confidential by: storing data on servers that are protected by high-end firewall systems, data will be encrypted so that information cannot be decoded, and we will not collect IP addresses. Every computer that communicates over the Internet is assigned an IP address that uniquely identifies the device. Data files, once downloaded, will be stored on Dr. Salazar's passwordprotected computer located in her locked office.

When we present or publish the results of this study, we will not use your name or other information that may identify you. The findings will be summarized and reported in group form. You will not be identified personally.

To further protect your privacy, this research is covered by a Certificate of Confidentiality from the National Institutes of Health. This Certificate will make sure we cannot be forced to share information that may identify you. The researchers will use the Certificate to resist any demands for information that would identify you, except for information from personnel of the United States Government that is used for other Federal projects. If you wish, you can share your information or involvement in this study with family and friends.

Version Date: July 31, 2018

| "Please check this box if you have read this section | on on the confidentiality of the research |
|---|---|
| study." | |

#### X. **Contact Persons:**

Contact Dr. Laura Salazar at 404-413-1396

- If you have questions about the study and your part in it
- If you have questions, concerns, or complaints about the research
- If you think you have been harmed by the study

Contact the GSU Office of Human Research Protections at 404-413-3500 or irb@gsu.edu

- If you have questions about your rights as a research participant
- If you have questions, concerns, or complaints about the research

| "Please check this box if you have read this section on the contact persons of the research |
|---|
| study." |

## Copy of Consent Form to Participant: XI.

Version Date: July 31, 2018

You can print a copy of this consent form to keep.

If you are willing to volunteer for this research please click on the "Continue" button.